CLINICAL TRIAL: NCT07041112
Title: Pharmacogenetic Observational Study Evaluating the Influence of Genetic Variants and Cardiometabolic Risk Factors on 10-Year Survival of Biologic Therapies in Patients With Cutaneous Psoriasis With or Without Psoriatic Arthritis
Brief Title: Ten-Year Biologic Drug Survival in Psoriasis: Role of Genetic and Cardiometabolic Predictors
Acronym: GENBIOPSO
Status: Completed | Type: Observational
Sponsor: Juan Ruano Ruiz (Other)
Collaborators: Hospital Universitario Reina Sofia de Cordoba (Other Government); Universidad de Córdoba (Other); Maimonides Institute for Biomedical Research of Cordoba (IMIBIC) (Unknown)
Responsible Party: Sponsor-Investigator, Juan Ruano Ruiz, Principal Investigator, IMIBIC-HURS, Córdoba, Spain, Maimónides Biomedical Research Institute of Córdoba
Organization: Maimónides Biomedical Research Institute of Córdoba (Other)
Other Study IDs: PSO-BIO-CSP-001; ICI1400136 (Other Grant/Funding Number: Instituto de Salud Carlos III (ISCIII), Spanish Ministry of Science, Innovation and Universities)
Record Dates: First submitted 2025-06-19; First posted 2025-06-27 (Actual); Last update posted 2025-06-27 (Actual); Status verified 2025-06

CONDITIONS: Psoriasis; Psoriatic Arthritis (PsA); Cardiovascular Risk Factors; Metabolic Syndrome (MetS); Drug Survival; Pharmacogenetics
Keywords: Biologic Therapy; Psoriasis Cohort; Genetic Variants; SNPs; Cytokines; Drug Durability; Real-World Data; Metabolic Biomarkers; Cardiometabolic Risk; Personalized Medicine; Inflammatory Skin Disease
MeSH Terms: conditions — Psoriasis; Arthritis, Psoriatic; Metabolic Syndrome; Dermatitis | interventions — Biological Therapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Peripheral blood samples were collected and stored for genomic DNA extraction. The retained biospecimens include EDTA-anticoagulated whole blood and plasma. DNA was used for genotyping of single nucleotide polymorphisms (SNPs) across 65 candidate genes related to psoriasis, metabolic syndrome, and cardiovascular risk. Plasma aliquots were preserved for cytokine, chemokine, and cardiometabolic biomarker profiling. All samples were coded and stored under standardized biobank conditions.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Psoriasis Cohort - Observational Follow-up: Adult patients with a confirmed diagnosis of plaque psoriasis, with or without psoriatic arthritis, who initiated biologic therapy between 2010 and 2020 at tertiary dermatology clinics in Spain. Participants were followed retrospectively for up to 10 years to assess treatment survival, safety, and disease outcomes. The study explores the influence of genetic variants (450 SNPs across 65 genes), cardiometabolic comorbidities, lifestyle factors, and circulating biomarkers (adipokines, cytokines, microparticles) on treatment durability and response. No interventions were assigned by protocol.
  Interventions: Drug: Biologic therapy for psoriasis

INTERVENTIONS:
Drug: Biologic therapy for psoriasis — Exposure to systemic biologic drugs for psoriasis, including TNF inhibitors (etanercept, adalimumab, infliximab, certolizumab), IL-12/23 inhibitors (ustekinumab), IL-17 inhibitors (secukinumab, ixekizumab, brodalumab), and IL-23 inhibitors (guselkumab, risankizumab, tildrakizumab). Treatments were prescribed as part of routine clinical care.
  Other Names: Anti-TNF, Anti-IL-12/23, Anti-IL-17, Anti-IL-23

SUMMARY:
This retrospective observational study aims to evaluate the long-term survival of biologic therapies in adult patients with moderate-to-severe cutaneous psoriasis, with or without psoriatic arthritis, over a period of up to 10 years. The study investigates the influence of clinical, metabolic, and genetic factors, including SNPs and metabolic syndrome components, on treatment durability. Data were obtained from a single-centre cohort treated in routine clinical practice. This analysis seeks to identify predictors of therapeutic response and to explore pharmacogenetic profiles that may inform personalized treatment strategies.

DETAILED DESCRIPTION:
This retrospective observational cohort study investigates the influence of clinical, anthropometric, lifestyle, cardiometabolic, immunological, and genetic factors on the long-term effectiveness and durability of biologic therapies in patients with moderate-to-severe plaque psoriasis, with or without psoriatic arthritis.

The study includes adult patients diagnosed with plaque psoriasis who initiated treatment with a biologic agent between 2011 and 2021 at a tertiary academic dermatology center. All subjects were systematically assessed through standardized procedures, and follow-up data were collected over a period of up to 10 years. The primary endpoint is biologic drug survival (time to discontinuation), while secondary endpoints include treatment response (PGA), presence of psoriatic arthritis, nail psoriasis, and family history of psoriasis.

Clinical and biomarker data collected at baseline included:

Anthropometric variables: body mass index (BMI), waist circumference.

Lifestyle indicators: Mediterranean diet adherence (MEDAS), physical activity frequency, smoking and alcohol habits, and perceived stress scale.

Cardiovascular and metabolic status: history and treatment of hypertension, type 2 diabetes mellitus, dyslipidemia, and metabolic syndrome, following ATP III/NCEP criteria.

Cardiometabolic biomarkers: leptin, adiponectin, insulin, lipoprotein(a), and HOMA-IR.

Inflammatory profile: a multiplex panel of cytokines and chemokines (including IL-1β, IL-6, IL-8, IL-17, IL-23, TNF-α, IFN-γ, MCP-1, IP-10).

Microparticles: circulating endothelial and platelet-derived microparticles quantified by flow cytometry.

Genotyping was performed using a custom array targeting 450 SNPs in 65 candidate genes previously associated with psoriasis susceptibility, systemic inflammation, and cardiometabolic risk (e.g., IL12B, IL23R, TNFAIP3, TRAF3IP2, HLA-C, CDKAL1, TCF7L2). Quality control included filtering by call rate, Hardy-Weinberg equilibrium, and minor allele frequency (MAF > 5%).

Data integration and quality assurance:

Clinical, laboratory, and genotyping data were integrated using unique patient identifiers.

A complete data dictionary was compiled, with defined variable sources, coding rules (e.g., WHO-ATC for drugs), and standard ranges.

Logical and range-based data checks were conducted. Variables with implausible values (e.g., negative survival time) were excluded or corrected.

A pre-specified imputation plan was applied to address missingness: median or mode imputation for clinical variables; multiple imputation for biomarkers where appropriate.

Variables were harmonized across data sources to ensure consistent definitions and temporal alignment.

All analyses adhered to a predefined statistical analysis plan.

Sample size and power: With over 800 patients and a median follow-up of 5+ years, the study has sufficient statistical power (>80%) to detect hazard ratios of ~1.5 for binary predictors with moderate prevalence (≥20%).

Statistical analysis:

Cox proportional hazards regression was used to assess the association between predictors and biologic drug survival.

Models were adjusted for potential confounders such as age, gender, and comorbidities.

Univariate models were conducted for each clinical and lifestyle variable, excluding SNPs, with false discovery rate (FDR) adjustment.

Stratified analyses were conducted by drug class (e.g., anti-TNF, anti-IL17, anti-IL12/23) and individual drug.

Pharmacogenetic analyses were conducted separately using additive models for each SNP, with interaction testing for cardiometabolic traits.

Results were summarized as hazard ratios (HR) with 95% confidence intervals and adjusted p-values.

All procedures followed STROBE guidelines for observational research. The study protocol was reviewed and approved by the Institutional Ethics Committee, and all patients provided written informed consent for biobanking and retrospective analysis of anonymized data.

This study aims to identify actionable clinical and genetic predictors of biologic therapy durability in real-world psoriasis, contributing to personalized treatment strategies and understanding of cardio-dermatologic interactions.

ELIGIBILITY:
Inclusion Criteria:

* Adults (≥18 years) diagnosed with moderate-to-severe cutaneous psoriasis.
* Initiation of treatment with a biologic agent between 2010 and 2020.
* Minimum follow-up of 12 months or until drug discontinuation.
* Availability of clinical and treatment data at baseline.
* Availability of at least one blood sample for biomarker/genetic analysis.
* Informed consent obtained for biobanking and genetic analyses.

Exclusion Criteria:

* Diagnosis of other chronic inflammatory skin diseases (e.g., atopic dermatitis, lupus).
* Concomitant participation in interventional clinical trials at baseline.
* Patients with incomplete treatment history or missing survival data.
* Systemic immunosuppressive therapy (e.g., cyclosporine, methotrexate) without biologics during the study period.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients (≥18 years) with moderate-to-severe cutaneous psoriasis, with or without psoriatic arthritis, who initiated treatment with biologic therapies at a tertiary dermatology center between 2010 and 2020. All participants had routine clinical follow-up and available biological samples for biomarker and genetic analyses.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Actual)
Dates: Start 2012-01-01 (Actual); Primary Completion 2023-03-01 (Actual); Study Completion 2024-06-01 (Actual)

PRIMARY OUTCOMES:
Drug survival at 10 years | Up to 10 years from treatment start
  Time from initiation of the biologic treatment to discontinuation for any cause (inefficacy, adverse events, remission, patient decision, etc.).

SECONDARY OUTCOMES:
Predictors of biologic drug discontinuation in patients with psoriasis | Up to 10 years from treatment initiation
  Clinical, metabolic, lifestyle and immunologic variables (including soluble cytokines, chemokines and microparticles) associated with biologic treatment discontinuation will be evaluated using multivariable Cox models.
Association between baseline soluble immune biomarkers and biologic drug survival | Up to 10 years from treatment initiation
  The association between baseline levels of cytokines, chemokines and other plasma-soluble biomarkers and long-term biologic drug survival will be assessed.
Genetic variants associated with baseline soluble immune biomarker levels | Baseline (pre-treatment)
  Genotyping data from 450 SNPs in 65 genes will be analyzed to identify variants associated with baseline levels of soluble cytokines, chemokines, and related immunometabolic markers.
Mediation of genetic effects on biologic survival by soluble immune biomarkers | From baseline to 10 years
  Mediation models will be used to evaluate whether baseline levels of soluble immune biomarkers explain, partially or fully, the effect of genetic variants on biologic drug survival.
Incidence of new-onset psoriatic arthritis (PsA) during follow-up | From baseline to 10 years
  The cumulative incidence of new PsA diagnosis will be recorded during follow-up among patients with cutaneous psoriasis initially free of PsA. Diagnosis will be confirmed by rheumatologists following CASPAR criteria.
Predictors of new-onset psoriatic arthritis during biologic treatment | From baseline to 10 years
  Baseline clinical, serological, genetic, and treatment-related factors associated with the risk of developing PsA during follow-up will be analyzed using Cox models and logistic regression.
Incidence and type of adverse events during biologic treatment | From baseline to 10 years
  Adverse events (AEs) reported during follow-up will be classified and recorded, including infections, cardiovascular events, malignancies, and other serious or treatment-related AEs.
Predictors of adverse events during biologic treatment | From baseline to 10 years
  Baseline clinical, metabolic, genetic and treatment-related variables will be analyzed to identify predictors of adverse events during treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Dermatology, Reina Sofia University Hospital, Córdoba, Córdoba, Spain

IPD SHARING:
Plan to Share IPD: Undecided
Individual participant data (IPD) will not be shared at this time. However, data sharing may be considered in the future once additional analyses are completed or if integration with other datasets is agreed upon as part of collaborative research efforts.

REFERENCES:
- [Background] Ruano J, Velez A, Casas E, Rodriguez-Martin A, Salido R, Isla-Tejera B, Espejo-Alvarez J, Gomez F, Jimenez-Puya R, Moreno-Gimenez JC. Factors influencing seasonal patterns of relapse in anti-TNF psoriatic responders after temporary drug discontinuation. J Eur Acad Dermatol Venereol. 2014 Apr;28(4):516-8. doi: 10.1111/jdv.12210. Epub 2013 Jul 11. No abstract available. PMID 23841941
- [Derived] de Luque J, Mochon-Jimenez C, Rivera-Ruiz I, Gay-Mimbrera J, Fuentes-Duculan J, Coats I, Aguilar-Luque M, Isla-Tejera B, Nieto AV, Galan-Gutierrez M, Lopez TL, Suarez-Farinas M, Krueger JG, Ruano J. A Functional Genetic Score in the ZMIZ1/TGF-beta/STAT Pathway Predicts Early Biologic Discontinuation in Psoriasis Patients Treated with Anti-TNF and Anti-IL12/23 Agents. Adv Ther. 2025 Dec;42(12):6030-6044. doi: 10.1007/s12325-025-03350-0. Epub 2025 Oct 6. PMID 41051639